CLINICAL TRIAL: NCT03119766
Title: Multicenter Double-blind Placebo-controlled Randomized Clinical Trial of Efficacy and Safety of Kolofort in the Treatment of Patients With Functional Dyspepsia
Brief Title: Clinical Trial of Efficacy and Safety of Kolofort in Functional Dyspepsia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-KOL-003
Record Dates: First submitted 2017-04-04; First posted 2017-04-19 (Actual); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2019-06

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kolofort (Experimental): Tablet for oral use. Dose per administration: 2 tablets. 2 tablets twice daily (4 tablets per day). The tablets should be held in the mouth until complete dissolution, without meal.
  Interventions: Drug: Kolofort
- Placebo (Placebo Comparator): Tablet for oral use. Dose per administration: 2 tablets. 2 tablets twice daily (4 tablets per day). The tablets should be held in the mouth until complete dissolution, without meal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kolofort — Oral administration
  Arms: Kolofort
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
Purpose of the study:

To obtain additional data on efficacy and safety of Kolofort in the treatment of patients with functional dyspepsia.

DETAILED DESCRIPTION:
Design: a multicenter double-blind placebo-controlled randomized clinical trial to evaluate the efficacy and safety of the study treatment.

The study will enroll the patients of both genders aged 18-45 years old with verified diagnosis of "functional dyspepsia" according to Rome-IV criteria and intensity of dyspeptic symptoms ≥ 6 according to GIS (Gastrointestinal symptom score).

At the screening visit 1 (Visit 1, from -14 to -1 days), after signing patient information sheet (informed consent form) to participate in the clinical trial, complaints and medical history are collected, an objective examination is performed. The investigator evaluates intensity of dyspeptic symptoms according to GIS. The patient undergoes an abdomen ultrasound examination, esophagogastroduodenoscopy (EGDS) , and diagnostic tests for Helicobacter pylori (H. pylori) infection. In case of the previous use of proton pump inhibitors, prokinetics, antispasmodics, antacids, bismuth drugs the investigator evaluates the possibility of canceling these drugs at least 7 days before the patient is randomized. For women of reproductive age, a pregnancy test is performed.

On the day of randomization (Visit 2, Day 0) collection of complaints and objective examination are carried out. The investigator evaluates the results of laboratory and instrumental research methods, the severity of dyspepsia symptoms on the GIS scale, registers changes in concomitant therapy.

If a patient meets all inclusion criteria and does not have any exclusion criteria, he/she is randomized into one of two groups: patients in Group 1 receive Kolofort for 8 weeks; patients in Group 2 - Placebo on the study drug regimen. The patient completes the Nepean Dyspepsia Index (NDI) and Quality of Life (SF-36) questionnaires.

The patient's treatment lasts for 8 weeks, during which 3 visits to the research center are carried out. At Visit 3 (Week 2 ± 3 days), complaints are collected, an objective examination of the patient is performed. The investigator monitors the prescribed and concomitant therapy, evaluates the safety of therapy and the degree of adherence to treatment (compliance). At visit 4 (week 4±3 days) and 5 (week 8±3 days) the investigator collects complaints, registers the physical examination data, monitors the prescribed and concomitant therapy, assesses the safety of the treatment and compliance. Questionnaires GIS, NDI are filled in.

Additionally, at Visit 5 the patient fills out the SF-36 scale, the investigator fills out the Clinical Global Impression-Efficacy Index (CGI-EI).

The patients will be allowed to take symptomatic therapy and medications for their co-morbidities during the study, except for the medicines listed in "Prohibited Concomitant Treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders aged 18-45 years old.
2. Diagnosis of functional dyspepsia established according to Rome-IV criteria (2016).
3. Severity of symptoms of dyspepsia ≥ 6 on the GIS scale.
4. Negative test result for H. pylori infection .
5. Availability of signed patient information sheet and informed consent form for participation in the clinical trial.
6. Patients who gave their consent to use reliable contraception during the study

Exclusion Criteria:

1. Organic diseases of the gastrointestinal tract (gastroesophageal reflux disease (GERD), peptic ulcer, chronic pancreatitis, cholelithiasis, hepatosis, hepatitis, hepatic cirrhosis, etc.)
2. Verified diagnosis of other functional GI diseases, i.e. biliary dyskinesia, irritable bowel syndrome, etc.
3. Discontinuation of proton pump inhibitors, prokinetics, antispasmodics, antacids, bismuth preparations less than 7 days before randomization.
4. H. pylori eradication within 2 months prior to enrollment.
5. Intestinal infection within 2 months prior to enrollment.
6. History/suspicion of oncology of any location.
7. Previously diagnosed cardiovascular diseases with functional class IV (according to the classification of the New-York Heart Association, 1964), hypothyroidism, diabetes mellitus, chronic renal disease С3-5, hepatic diseases with portal hypertension and/or signs of severe decompensation of function (> 6 points according to the Child-Pugh classification).
8. Any other severe comorbidity that, in the opinion of the investigator, may affect patient participation in the clinical trial.
9. Allergy/intolerance intolerances to any of the components of the study drugs.
10. Pregnancy, breast-feeding.
11. Patients who, from the investigator's point of view, will not comply with the observation requirements of the study or adhere to study drug dosing regimens.
12. Scheduled hospitalization during the study for any diagnostic or therapeutic procedures.
13. Use of drugs or alcohol (more than 2 alcohol units daily), presence of mental diseases.
14. Use of any medications specified in the "Prohibited Concomitant Treatment" within 1 month prior to inclusion in the study.
15. Participation in other clinical trials in the previous 3 months.
16. Patients who are related to any of the on-site research personnel directly involved in the conduct of the trial or are an immediate relative of the study investigator. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
17. Patients who work for MATERIA MEDICA HOLDING (i.e. the company's employees, temporary contract workers, appointed officials responsible for carrying out the research or immediate relatives of the aforementioned).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 370 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- Russia (31):
  - South Ural State University, Chelyabinsk
  - Ivanovo Clinical Hospital named after Kuvaev, Ivanovo
  - State budget institution of health care of the Moscow region "Krasnogorsk city hospital №1", Krasnogorsk
  - The State Budgetary Healthcare Institution of Moscow The Moscow Clinical Scientific and Practical Center of the Moscow City Health Department, Moscow
  - Federal State Budgetary Institution Federal Research and Clinical Center for Specialized Medical Assistance and Medical Technologies of the Federal Medical Biological Agency of Russia, Moscow
  - The Federal State Budgetary Healthcare Institution The Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - The State Budget Educational institution of High Professional Training I.M. Sechenov First Moscow State Medical University of Ministry of Health Care of the Russian Federation, Moscow
  - National Medical Research Center for Rehabilitation and Health Resort, Moscow
  - State Budgetary Healthcare Institution of Moscow "City Clinical Hospital No. 51 of the Moscow City Health Department", Moscow
  - Federal State Budgetary Educational Institution of the Higher Education "A.I. Yevdokimov Moscow State University of Medicine and Dentistry" of the Ministry of Healthcare of the Russian Federation, Moscow
  - Federal State Budgetary Institution "Polyclinic No. 3" of the Administration of the President of the Russian Federation, Moscow
  - Private Healthcare Institution "The Road Clinical Hospital at the Nizhny Novgorod station of the open joint-stock company" Russian Railways ", Nizhny Novgorod
  - Novosibirsk State Medical University, Novosibirsk
  - State budgetary healthcare institution of the Moscow region "Podolsk City Clinical Hospital No. 3", Podol’sk
  - State Autonomous Healthcare Institution of the Moscow Region "Central City Clinical Hospital in Reutov", Reutov
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic №38", Saint Petersburg
  - State budget institution of higher education "North-Western State Medical University named after I.I Mechnikov" under the Ministry of Public Health of the Russian Federation, Saint Petersburg
  - City Mariinsky Hospital, Saint Petersburg
  - Federal state budget military educational institution of higher professional education "Military Medical Academy named after S.Kirov" of the Ministry of Defense of the Russian Federation, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Hospital of the Holy Martyr Elizabeth", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Hospital No. 26", Saint Petersburg
  - Limited Liability Company Gastroenterologichesky Center Expert, Saint Petersburg
  - Samara City Hospital #4, Samara
  - LLC Medical company "Hepatologist", Samara
  - Saratov State Medical University named after V. I. Razumovsky, Saratov
  - Saratov City Clinical Hospital #5, Saratov
  - St. Petersburg State Budgetary Institution "City Hospital No. 40 in the Kurortny District", Sestroretsk
  - Stavropol Regional Clinical Consultative and Diagnostic Center, Stavropol
  - State Healthcare Institution Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - State Autonomous Healthcare Institution of the Yaroslavl Region "N.V. Clinical Emergency Hospital Solovyov ", Yaroslavl
  - Municipal Budgetary Institution "Central City Hospital No. 7", Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 370 patients were enrolled in the study and signed informed consent. After undergoing screening procedures, 61 patients were excluded by the investigators because they did not meet the inclusion criteria, or they had non-inclusion criteria. 309 patients were randomized into two groups - 151 into Kolofort group and 158 into Placebo group.
Period: Overall Study
Arm/Group | Kolofort | Placebo
Started | 151 | 158
Completed | 151 | 158
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study will enroll the subjects of either gender aged 18-45 years old with verified diagnosis of "functional dyspepsia" according to Rome-IV criteria, intensity of dyspeptic symptoms ≥ 6 according to GIS and negative H. pylori test.
Groups:
- Total: Total of all reporting groups
Arm/Group | Kolofort | Placebo | Total
Number analyzed (Participants) | 151 | 158 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (7.7) | 29.7 (7.9) | 30.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 110 | 215
  Male | 46 | 48 | 94
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 151 | 158 | 309

OUTCOME MEASURES:

1. Primary Outcome: Changes in Severity of Functional Dyspepsia Symptoms
Description: Changes in severity of functional dyspepsia symptoms due to GIS score (Gastrointestinal symptom score) at week 8 from the start of study therapy. The GIS scale includes 10 subscales (symptoms), the severity of each one was evaluated from 0 to 4 points (by Lickert scale).For example, the absence of the mentioned symptom is classified as "0". The most severe is classified as "4".
  The all 10 subscales were combined to compute a total score. So the total range is a sum of all subscales.The total score is in range from 0 till 40. So the minimum value is 0, the maximum is 40.
Time Frame: On baseline, after 4 and 8 weeks of the treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kolofort | Placebo
Number analyzed (Participants) | 151 | 158
score on a scale
  Baseline score | 10.1 (3.1) | 10.0 (3.9)
  Score after 4 weeks | 5.1 (3.0) | 5.2 (3.0)
  Score after 8 weeks | 2.9 (2.5) | 3.7 (3.6)
  "Baseline minus 8 weeks" score difference | 7.2 (3.3) | 6.3 (4.6)
Statistical Analysis 1: Comparison: Kolofort vs Placebo; Mean changes of GIS scores after 8 weeks of treatment were compared; Test type: Superiority; p = 0.041, ANOVA; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [0.04 to 1.85] — Results are presented as estimated differences of Least Squares Means according to ANOVA model
Statistical Analysis 2: Comparison: Kolofort vs Placebo; Mean changes of GIS scores after 8 weeks of treatment were compared. Influence of between center variation was estimated; Test type: Superiority; p = 0.041, Mixed Models Analysis; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [0.04 to 1.74] — Fixed factor "Treatment" and random factor "research center" were used in mixed model. Difference in mean changes between groups was estimeted

2. Secondary Outcome: Percentage of Patients With a Decrease in the Severity of FD Symptoms
Description: Percentage of patients with a decrease in the severity of FD symptoms on the GIS scale after 8 weeks from the start of study therapy. The GIS scale is composed of 10 points evaluating the extent of manifestation of a wide range of gastroenterological symptoms. The intensity of clinical symptoms will be evaluated based on a 5-point Likert scale from 0 to 4 where 0 = no, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe).
Time Frame: After 8 weeks of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Kolofort | Placebo
Number analyzed (Participants) | 151 | 158
Participants
  Reduction ≥ 1 point | 150 | 151
  Reduction ≥ 2 points | 145 | 141
  Reduction ≥ 3 points | 138 | 134
  Reduction ≥ 4 points | 133 | 125
  Reduction ≥ 5 points | 121 | 114
Statistical Analysis 1: Comparison: Kolofort vs Placebo; Test for comparison percentage of patients with reduction ≥ 1 point; Test type: Superiority; p = 0.067, Fisher Exact
Statistical Analysis 2: Comparison: Kolofort vs Placebo; Test for comparison percentage of patients with reduction ≥ 2 points; Test type: Superiority; p = 0.029, Fisher Exact
Statistical Analysis 3: Comparison: Kolofort vs Placebo; Test for comparison percentage of patients with reduction ≥ 3 points; Test type: Superiority; p = 0.082, Fisher Exact
Statistical Analysis 4: Comparison: Kolofort vs Placebo; Test for comparison percentage of patients with reduction ≥ 4 points; Test type: Superiority; p = 0.046, Fisher Exact
Statistical Analysis 5: Comparison: Kolofort vs Placebo; Test for comparison percentage of patients with reduction ≥ 5 points; Test type: Superiority; p = 0.111, Fisher Exact

3. Secondary Outcome: Change in the Severity of the Functional Dyspepsia Index NDI (Nepean Dyspepsia Index)
Description: Change in the severity of the functional dyspepsia index NDI (Nepean dyspepsia index) after 8 weeks from the start of the study therapy. The NDI questionnaire involves the patient's self-assessment of various manifestations of the disease and how much FD affects his life. The range of possible fluctuations in the total score of the Nepean dyspepsia index is from 10 to 50.
  The scale consists of 10 questions. Each section corresponds to 5 answer options (the lower score is 1, the highest is 5), reflecting the gradation of the severity of the symptom and coded according to the increase in the severity of the symptom or the loss of the ability to perform a certain task in the framework of daily activities. The minimum value is 10, the maximum value is 50. The higher score represents the worst outcome.
Time Frame: On baseline, after 4 and 8 weeks of the treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kolofort | Placebo
Number analyzed (Participants) | 151 | 158
units on a scale
  Baseline | 23.5 (7.0) | 23.5 (6.9)
  After 4 weeks | 17.1 (5.6) | 17.0 (6.0)
  After 8 weeks | 14.4 (5.1) | 14.9 (6.0)
  "Baseline minus 8 weeks" score difference | 9.1 (7.1) | 8.5 (6.6)
Statistical Analysis 1: Comparison: Kolofort vs Placebo; Mean changes of NDI scores after 8 weeks of treatment were compared; Test type: Superiority; p = 0.435, ANOVA; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.93 to 2.15] — Results are presented as estimated differences of Least Squares Means according to ANOVA model

4. Secondary Outcome: Changes in the Quality of Life of Patients on the SF-36 (Short Form-36) Health Survey Scale
Description: The scale reflects the general well-being of a person, which is affected by the state of health, and consists of 11 questions. In the composition of the SF-36 dedicated 8 sections:1. Physical functioning,2. Role (physical) functioning 3. Pain.4. General health.5. Vitality.6. Social functioning.7. Emotional functioning. 8. Psychological health.The sections of the scale are combined into 2 total dimensions - the physical component of health (1-4 questions) and mental (5-8 questions). Subscales (questions 1-4) were summed to provide the information about the physical component, subscales (questions 5-8) - about the mental component. Each scale ranges from 0 to 100 so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
Time Frame: On baseline and after 8 weeks of the treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kolofort | Placebo
Number analyzed (Participants) | 151 | 158
score on a scale
  Baseline (physical score) | 49.9 (7.8) | 49.4 (7.7)
  After 8 weeks (physical score) | 56.3 (6.5) | 56.2 (6.3)
  "Baseline minus 8 weeks" score difference (physical score) | 6.4 (7.5) | 6.8 (7.0)
  Baseline (mental score) | 33.6 (5.7) | 34.0 (6.1)
  After 8 weeks (mental score) | 37.1 (4.5) | 36.9 (4.9)
  "Baseline minus 8 weeks" score difference (mental score) | 3.5 (6.3) | 2.9 (6.6)
Statistical Analysis 1: Comparison: Kolofort vs Placebo; Mean changes of SF-36 scores (physical health domain) after 8 weeks of treatment were compared; Test type: Superiority; p = 0.655, ANOVA; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-2.00 to 1.26] — Results are presented as estimated differences of Least Squares Means according to ANOVA model
Statistical Analysis 2: Comparison: Kolofort vs Placebo; Mean changes of SF-36 scores (mental health domain) after 8 weeks of treatment were compared; Test type: Superiority; p = 0.375, ANOVA; Median Difference (Final Values) = 0.65, 95% CI 2-sided [-0.79 to 2.10]

5. Secondary Outcome: Percentage of Patients Terminating the Study Early
Description: Percentage of patients terminating the study early due to lack of efficacy of the study therapy. Lack of efficacy of the study therapy is defined as retention or progression of the symptoms of functional dyspepsia resulting in prescription of the products for FD therapy (proton pump inhibitors, prokinetics, spasmolytics).
Time Frame: in 8 weeks of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Kolofort | Placebo
Number analyzed (Participants) | 151 | 158
Participants | 0 | 1
Statistical Analysis 1: Comparison: Kolofort vs Placebo; Test type: Superiority; p = 1, Fisher Exact

6. Secondary Outcome: Indicators of Therapeutic and Side Effects, Efficacy Index on CGI-EI (Clinical Global Impression-Efficacy Index) Scale
Description: Indicators of therapeutic and side effects, efficacy index on the scale of the general clinical impression CGI-EI (Clinical Global Impression Scale - Efficacy Index) after 8 weeks from the start of study therapy. Clinical Global Impression Efficacy Index (CGI-EI) will be filled by the investigator at the final Visit 5 (Week 8±3 days). Evaluation of the response to treatment should take into account both therapeutic efficacy and treatment-related side effects. Side effects value from 1 to 4. Therapeutic effect value as 0,4,8 or 12 points. The efficacy index is a sum. The minimum value is 1, the maximum value is 16. A lower score on the scales is the best outcome.
Time Frame: After 8 weeks of the treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kolofort | Placebo
Number analyzed (Participants) | 151 | 158
units on a scale
  Side effects | 1.09 (0.31) | 1.04 (0.19)
  Therapeutic effect | 2.67 (2.96) | 3.33 (3.49)
  Efficacy index | 3.76 (2.98) | 4.37 (3.51)
Statistical Analysis 1: Comparison: Kolofort vs Placebo; Side effects analysis; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Kolofort vs Placebo; Therapeutic effect; Test type: Superiority; p = 0.139, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Kolofort vs Placebo; Efficacy index analysis; Test type: Superiority; p = 0.251, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the treatment period - 8 weeks (start after taking the first dose of the study drug, during the entire period of the study therapy and within 24 hours after the last dose of the study drug).
Arm/Group | Kolofort | Placebo
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/158
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/158
Other Adverse Events (participants affected / at risk) | 13/151 | 12/158
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kolofort (N=151) | Placebo (N=158)
Hyperkinesia gastrointestinal intestinal tract (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
ARVI (Infections and infestations) | 2 (2) | 1 (1) — Upper respiratory tract infection
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pain in the oropharynx (oropharyngeal)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) — General weakness
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03119766/Prot_SAP_000.pdf